CLINICAL TRIAL: NCT03467282
Title: Effect of Probiotic Supplementation in Nonalcoholic Steatohepatitis Patients: Randomized Clinical Trial - PROBILIVER TRIAL
Brief Title: Probiotics in NASH Patients - PROBILIVER TRIAL
Acronym: NASH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 160438
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): 1g probiotic mix (twice day): Lactobacillus acidophilus 1x109 CFU + Bifidobacterium lactis 1x109 CFU + Lactobacillus rhamnosus 1x109 CFU + Lactobacillus paracasei 1x109 CFU
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): 1g polydextrose/maltodextrin - twice day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — 1g probiotic mix (twice day): Lactobacillus acidophilus 1x109 CFU + Bifidobacterium lactis 1x109 CFU + Lactobacillus rhamnosus 1x109 CFU + Lactobacillus paracasei 1x109 CFU
  Arms: Probiotic
Dietary Supplement: Placebo — 1g polydextrose/maltodextrin - twice day
  Arms: Placebo

SUMMARY:
Non-alcoholic Fatty Liver Disease (NAFLD) is characterized by excessive accumulation of lipids in hepatocytes, not associated with alcohol consumption and ranges from hepatic steatosis to steatohepatitis, a form that can progress to cirrhosis or hepatocarcinoma, and is considered a liver manifestation of the metabolic syndrome (MetS). The disease occurs in 16 - 30% of the general population, but can reach up to 90% of obese individuals. Changes in lifestyle, including weight loss and physical activity are indicated with first choices for improvement of the liver condition.

Recently the relationship between obesity, diabetes, MetS and NAFLD with intestinal microbiota has also been suggested in the development and progression of liver disease, since it is related to hepatic steatosis and inflammation. In this sense, this work aims to evaluate the effects of probiotic supplementation on intestinal microbiota modulation, degree of hepatic fibrosis and steatosis, inflammation and body composition.

DETAILED DESCRIPTION:
In this randomized clinical trial (RCT) will include adult outpatients linked to the Gastroenterology Service of the Hospital de Clínicas de Porto Alegre (Hospital of Clinics of Porto Alegre-HCPA) -Brazil with diagnosis of NAFLD confirmed by biopsy and transient elastography. Patients who are cirrhotic, pregnant, co-infected or who have Chronic Kidney Disease will not be included. All patients, after signing the Written Informed Consent Form, will undergo a complete anamnesis to investigate alcohol consumption (AUDIT, Alcohol Use Disorders Identification Test), smoking, previous history, medications in use, food consumption assessment (through a 3-day food record), physical activity level and physical and functional capacity (International Physical Activity Questionnaire, sit-to-stand test, unipodal, walk test and dynamometry), body composition (Electrical bioimpedance, dual energy x-ray absorptiometry (DEXA), anthropometric measurements), cardiovascular risk (Framingham Score and Atherosclerotic Cardiovascular Disease - ASCVD), biochemical parameters for assessment of inflammatory status [C-reactive protein (CRP), toll-like receptor 4 (TLR4)], lipid profile (total cholesterol, HDL, LDL, triglycerides), hepatic function [cytokeratin-18 (CK18), aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyltransferase (GGT), bilirubin, alkaline phosphatase], as well as blood glucose level , insulin, albumin, creatinine and complete blood count and even assessment of gut microbiota (patients will be provided with a kit for collecting feces and from the extraction of DNA from stool samples, after which a metagenomic analysis will be performed). These procedures will be performed at baseline and repeated after 24 weeks (at the end of the study). Through the of process of randomization (randomization.com), the patients will be allocated to receive treatment A or B. As for patients and researchers involved both are blinded (double-blind study). The intervention consists of treatment with probiotic mix (Lactobacillus acidophilus 1x109 colony-forming unit (CFU) + Bifidobacterium lactis 1x109 CFU + Lactobacillus rhamnosus 1x109 CFU + Lactobacillus paracasei 1x109 CFU) and the placebo identical in characteristics and packaging (polydextrose/maltodextrin). Patients will be instructed to consume 2 sachets/day during 24 weeks. Patients will be instructed to report any symptoms or para effects related to the use of sachets and adherence control will be carried out through the patient's notes on a form provided and also by checking the number of sachets.

ELIGIBILITY:
Inclusion Criteria:

* adult outpatient with diagnostic of NAFLD

Exclusion Criteria:

* HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV) infected patients
* significant intake of alcohol
* cirrhosis,
* pregnant women,
* transplanted patients,
* intake of supplements or foods containing probiotics,
* immunosuppressants, antibiotics, corticosteroids, valproic acid and amiodarone,
* other chronic inflammatory diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
hepatic fibrosis | 24 weeks
  change in the degree of fibrosis by hepatic elastography and scores
cardiovascular risk | 24 weeks
  change in scores and sistemic markers

SECONDARY OUTCOMES:
diversity of gut microbiota | 24 weeks
  by metagenomics from faecal samples
inflammation by TLR4 expression | 24 weeks
  by ELISA
inflammation by CK18 expression | 24 weeks
  by ELISA
inflammation by serum C-reactive protein | 24 weeks
  by nephelometry
metabolic syndrome | 24 weeks
  reduce in number of metabolic syndrome components
change in body composition by DEXA | 24 weeks
  densitometer GE Medical Systems Lunar Prodigy
body composition by bioimpedance | 24 weeks
  by change in phase angle
change in hand grip strength | 24 weeks
  by manual dynamometry
change in physical ability | 24 weeks
  by walk speed test
change in the parameters of sarcopenia by serum myostatin | 24 weeks
  by ELISA
change in the parameters of sarcopenia by serum testosterone | 24 weeks
  by electrochemiluminescence

CONTACTS AND LOCATIONS:
Overall Officials: Valesca Dall Alba, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barcelos STA, Silva-Sperb AS, Moraes HA, Longo L, de Moura BC, Michalczuk MT, Uribe-Cruz C, Cerski CTS, da Silveira TR, Dall'Alba V, Alvares-da-Silva MR. Oral 24-week probiotics supplementation did not decrease cardiovascular risk markers in patients with biopsy proven NASH: A double-blind placebo-controlled randomized study. Ann Hepatol. 2023 Jan-Feb;28(1):100769. doi: 10.1016/j.aohep.2022.100769. Epub 2022 Oct 8. PMID 36216309
- [Derived] Silva-Sperb AS, Moraes HA, de Moura BC, Alves BC, Bruch-Bertani JP, Azevedo VZ, Dall'Alba V. Effect of probiotic supplementation in nonalcoholic steatohepatitis patients: PROBILIVER TRIAL protocol. Trials. 2019 Oct 10;20(1):580. doi: 10.1186/s13063-019-3679-7. PMID 31601229